CLINICAL TRIAL: NCT07014839
Title: Biomarkers Predicting Postimplantation Syndrome After Endovascular Aortic Repair (EVAR) and Thoracic Endovascular Aortic Repair (TEVAR)
Brief Title: Post-Implantation Syndrome and Laboratory Markers Following EVAR and TEVAR
Acronym: PIS and EVAR
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ümit arslan, Associate Professor, Ataturk University
Other Study IDs: UA_ES_01
Record Dates: First submitted 2025-05-12; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Postimplantation Syndrome; Endovascular Abdominal Aortic Aneurysm Repair (EVAR); Thoracic Endovascular Aortic Repair
Keywords: Postimplantation Syndrome; Endovascular repair of aortic aneurysms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Implantation Syndrome: Lab Trends after EVAR/TEVAR: This cohort includes patients who underwent endovascular aneurysm repair (EVAR) or thoracic endovascular aortic repair (TEVAR). The study investigates the occurrence of post-implantation syndrome (PIS) and its association with early postoperative laboratory markers, including interleukin-6 (IL-6), neutrophil-to-lymphocyte ratio (NLR), leukocyte count, C-reactive protein (CRP), and procalcitonin levels. No additional pharmacologic or procedural interventions were applied beyond standard perioperative care.
  Interventions: Procedure: Endovascular Aortic Intervention

INTERVENTIONS:
Procedure: Endovascular Aortic Intervention — This intervention involves EVAR or TEVAR for the treatment of abdominal or thoracic aortic aneurysms, respectively. The procedures were performed using commercially available stent-grafts via a transfemoral approach under standard perioperative protocols. The study specifically focuses on the systemic inflammatory response following these interventions, with close monitoring of laboratory parameters including IL-6, neutrophil-to-lymphocyte ratio (NLR), CRP, leukocyte count, and procalcitonin during the early postoperative period. No adjunctive anti-inflammatory or immunomodulatory therapies were administered.

SUMMARY:
The aim of this observational study is to investigate the relationship between postimplantation syndrome (PIS) and laboratory inflammatory parameters following endovascular aortic repair (EVAR/TEVAR). PIS is a systemic inflammatory response that may occur after EVAR or TEVAR and lacks a standardized clinical definition. This study seeks to determine whether specific laboratory biomarkers-particularly white blood cell count, C-reactive protein (CRP), interleukin levels, and neutrophil-to-lymphocyte ratio (NLR)-can serve as reliable indicators for the diagnosis and assessment of PIS.

DETAILED DESCRIPTION:
Endovascular repair of thoracic and abdominal aortic aneurysms (EVAR/TEVAR) has become a preferred alternative to open surgical repair due to its association with reduced perioperative morbidity and mortality. However, a notable proportion of patients undergoing these procedures may develop postimplantation syndrome (PIS), a systemic inflammatory response first described in 1999. Despite its clinical relevance, PIS remains poorly defined, with varying diagnostic criteria across the literature.

PIS is typically characterized by postoperative fever, fatigue, and an increase in inflammatory markers such as white blood cell (WBC) count, C-reactive protein (CRP), and interleukin-6 (IL-6). The neutrophil-to-lymphocyte ratio (NLR), a readily obtainable marker from complete blood count tests, has also gained attention as a reliable indicator of systemic inflammation. In contrast, procalcitonin levels in PIS patients often remain within normal limits, helping differentiate PIS from bacterial infections.

In this prospective observational study, 200 patients undergoing elective EVAR or TEVAR procedures under general anesthesia were included. All procedures were performed via bilateral femoral artery access using open femoral incisions. Patients were followed postoperatively and assessed for the development of PIS based on clinical and laboratory parameters.

Body temperature was measured at regular intervals, and inflammatory markers-including CRP, WBC count, IL-6, NLR, and procalcitonin-were recorded preoperatively and at 24, 48, and 72 hours postoperatively. PIS was defined as the presence of fever (>38°C) in association with elevated CRP and/or leukocytosis, in the absence of any clinical or microbiological evidence of infection.

Preliminary results showed that patients who developed PIS had significantly higher postoperative levels of WBC, CRP, IL-6, and NLR, while procalcitonin levels remained normal, supporting a non-infectious inflammatory etiology. Imaging and laboratory evaluations ruled out alternative sources of infection. No significant differences were observed in operative time or graft type between patients with and without PIS.

All data were collected prospectively and analyzed using the SPSS statistical software. The study aims to clarify the diagnostic criteria of PIS by identifying specific laboratory biomarkers that can reliably differentiate PIS from other postoperative complications, particularly infection. Furthermore, by better understanding the inflammatory response following EVAR/TEVAR, the study may contribute to improved postoperative management strategies.

ELIGIBILITY:
Inclusion Criteria

* Patients aged ≥18 years
* Undergoing elective EVAR or TEVAR for abdominal or thoracic aortic aneurysm
* Ability to provide informed consent
* Availability of baseline and follow-up laboratory data (including IL-6, NLR, CRP, leukocyte count, procalcitonin, etc.)

Exclusion Criteria

* Evidence of active infection at the time of procedure
* Known autoimmune or inflammatory disease (e.g., rheumatoid arthritis, lupus)
* Current use of immunosuppressive or anti-inflammatory therapy
* Malignancy under active treatment
* End-stage renal or hepatic failure
* Emergency or ruptured aneurysm repair
* Incomplete postoperative laboratory data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) who underwent elective endovascular aneurysm repair (EVAR) or thoracic endovascular aortic repair (TEVAR) for abdominal or thoracic aortic aneurysms at a single tertiary care center. All participants had available pre- and postoperative laboratory data necessary for the evaluation of post-implantation syndrome and inflammatory biomarkers.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Postimplantation Syndrome (PIS) Incidence | 0-8 days
  PIS is defined as the presence of fever (>38°C) without an identifiable source of infection, accompanied by leukocytosis (white blood cell count >12,000/mm³) and/or elevated C-reactive protein (CRP >7 mg/L). The incidence rate of PIS will be calculated based on the number of patients meeting these diagnostic criteria following EVAR or TEVAR procedures.
  Unit of Measure:
  Percentage of participants with PIS (%)

SECONDARY OUTCOMES:
C-reactive Protein (CRP) Level | within first 72 hours postoperatively
  Serum CRP levels will be measured preoperatively and within 72 hours postoperatively. CRP values >7 mg/L will be considered elevated and potentially supportive of PIS diagnosis.
  Unit of Measure:
  mg/L
White Blood Cell (WBC) Count | within first 72 hours postoperatively
  Total leukocyte count will be assessed preoperatively and within 72 hours postoperatively. Values >12,000/mm³ will be considered elevated.
  Unit of Measure:
  10³ cells/μL
Interleukin-6 (IL-6) Level | within first 72 hours postoperatively
  Plasma IL-6 concentration will be measured preoperatively and within 72 hours postoperatively. IL-6 levels >7 ng/mL will be considered indicative of systemic inflammation.
  Unit of Measure:
  ng/mL
Neutrophil-to-Lymphocyte Ratio (NLR) | within first 72 hours postoperatively
  Neutrophil-to-Lymphocyte Ratio (NLR)
  Description:
  NLR will be calculated from the differential leukocyte count. A value >4 will be used as a cut-off indicating systemic inflammatory response.
  Unit of Measure:
  Unitless (ratio)
Procalcitonin (PCT) Level | within first 72 hours postoperatively
  Serum procalcitonin levels will be evaluated preoperatively and within 72 hours postoperatively. PCT <1 ng/mL will be considered as non-specific for bacterial infection but still relevant in inflammatory profiling.
  Unit of Measure:
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: umit arslan, Principal Investigator — Ataturk University
Locations (2):
- Turkey (Türkiye) (2):
  - Atatürk University, Erzurum
  - Ataturk University, Erzurum

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made publicly available due to institutional policies and the potential for overlapping use of the same dataset by other researchers within the institution. However, data may be shared upon reasonable request, provided that appropriate ethical approvals and data-sharing agreements are in place

REFERENCES:
- [Result] D'Oria M, Manoranjithan S, Scoville C, Vogel TR, Cheung S, Calvagna C, Lepidi S, Bath J. Systematic review of risk factors and outcomes of post-implantation syndrome following endovascular aortic repair. J Vasc Surg. 2024 May;79(5):1240-1250.e4. doi: 10.1016/j.jvs.2023.12.029. Epub 2023 Dec 18. PMID 38122858

DOCUMENTS (1):
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT07014839/ICF_000.pdf